CLINICAL TRIAL: NCT07032402
Title: The Effect of the Use of ABÖS-M App Developed for Mothers With Newborn Babies on Knowledge, Skills and Self-Efficacy Levels: Randomized Controlled Study
Brief Title: The Effect of the Use of Mobile App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 04012024
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Sudden Infant Death Syndrome
Keywords: Sudden Infant Death Syndrome; Mobile Applications; Neonatal Nursing; Randomized Controlled Trial
MeSH Terms: conditions — Sudden Infant Death | interventions — Educational Status; Counseling; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Group I (Experimental): Behavioral and Counseling
  Interventions: Behavioral: Education and Counseling
- Control: Group II (Other): Standard Care
  Interventions: Other: Standard Care

INTERVENTIONS:
Behavioral: Education and Counseling — Mothers who consent will have the ABÖS-M App installed on their smartphones and will create a personal login. Researchers will provide brief training on how to use the app. The intervention consists of four educational modules designed with individualized and gamified content. Mothers are expected to complete all modules within two weeks. The app monitors their progress and provides automated feedback based on their performance, encouraging mothers to review topics if needed. Weekly WhatsApp reminders will be sent to promote app engagement, and researchers will track login frequency and usage time. Mothers who fail to complete the modules within the specified timeframe will be excluded from the study. Participants will also be asked to fill out a daily care diary throughout the intervention period.
  Arms: Experimental: Group I
Other: Standard Care — After obtaining written and verbal consent, the ABÖS-M App will be installed on their smartphones, and researchers will provide face-to-face instructions on its basic use. Mothers in the control group will receive routine newborn care education provided by clinical nurses, which includes non-standardized safe sleep information typically given before hospital discharge. No structured or individualized training will be provided by the researchers during the study period. For one month, control group participants will have limited access to certain app features, including the "About Us" section, care diary, and assessment tools. Mothers will be asked to complete the care diary daily, and researchers will send regular reminders.
  Arms: Control: Group II

SUMMARY:
This randomized controlled trial aims to evaluate the effect of using the ABÖS-M mobile application, developed for mothers with newborns, on maternal knowledge, care skills, and self-efficacy levels related to Sudden Infant Death Syndrome (SIDS).

DETAILED DESCRIPTION:
Informing and raising parental awareness on Sudden Infant Death Syndrome (SIDS) and safe sleeping practices is crucial for promoting public health. This study aims to inform mothers about the risk factors involved in SIDS and encourage them to maintain a safe sleeping environment to safeguard their babies. As part of this study, the investigators intend to create a personalised, gamified mobile application training programme for mothers called the ABÖS-M App. Our main objective is to analyse the impact of ABÖS-M App on the knowledge, skills, and self-efficacy levels of mothers. To date, the investigators have not found any randomised controlled studies in Turkey that aim to prevent SIDS. Our study was designed as a single-centre, follow-up, single-blind, randomised controlled trial. The study was designed to include 25 mothers each in the intervention and control groups. The data was collected through a set of forms including the Information Form for Infants and Parents, the Sudden Infant Death Syndrome Knowledge Level Self-Assessment Form, the Sudden Infant Death Syndrome Care Skills Form, and the General Self-Efficacy Scale. Data analysis will be conducted using the Statistical Package for Social Science (SPSS v.23) software licensed by Akdeniz University. Repeated measures will be employed in the investigation to compare the measurements and scores between the intervention and control groups. Spearman correlation analysis will be utilised to evaluate the degree of relationship between the measurements. A significance level of p<0.05 will be considered. Additionally, the effect size of the study will be computed. Consequently, it is anticipated that the ABÖS-M App will enhance the knowledge, skills and self-efficacy levels of the mothers by the end of this project.

ELIGIBILITY:
Inclusion Criteria:

* Mothers with a healthy newborn baby,
* Mothers who have not experienced any previous child loss,
* Mothers with at least a primary school education,
* Mothers who own a smartphone with mobile internet access,
* Mothers who speak Turkish, are able to understand written and spoken information, follow instructions, and have no communication barriers,
* Mothers who voluntarily agree to participate in the study.

Exclusion Criteria:

* Mothers with postpartum depression,
* Mothers who do not complete the educational program within 15 days,
* Mothers who request withdrawal from the study at any stage.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Knowledge | baseline (first assessment)
  The Sudden Infant Death Syndrome Knowledge Self-Assessment Form was developed by the researchers based on the safe sleep recommendations of the American Academy of Pediatrics and the relevant literature to assess mothers' knowledge levels and caregiving skills related to the causes, risk factors, and preventive interventions for Sudden Infant Death Syndrome. The form consists of a total of 28 items: 3 items assessing general knowledge about SIDS, 15 items evaluating SIDS risk factors, and 10 items evaluating protective factors. The scores obtainable from the form range from 0 to 27. An increase in the score indicates a higher level of knowledge.
Knowledge | 2 weeks after from baseline
  The Sudden Infant Death Syndrome Knowledge Self-Assessment Form was developed by the researchers based on the safe sleep recommendations of the American Academy of Pediatrics and the relevant literature to assess mothers' knowledge levels and caregiving skills related to the causes, risk factors, and preventive interventions for Sudden Infant Death Syndrome. The form consists of a total of 28 items: 3 items assessing general knowledge about SIDS, 15 items evaluating SIDS risk factors, and 10 items evaluating protective factors. The scores obtainable from the form range from 0 to 27. An increase in the score indicates a higher level of knowledge.
Knowledge | at the end of the invervention program (4 weeks after from baseline)
  The Sudden Infant Death Syndrome Knowledge Self-Assessment Form was developed by the researchers based on the safe sleep recommendations of the American Academy of Pediatrics and the relevant literature to assess mothers' knowledge levels and caregiving skills related to the causes, risk factors, and preventive interventions for Sudden Infant Death Syndrome. The form consists of a total of 28 items: 3 items assessing general knowledge about SIDS, 15 items evaluating SIDS risk factors, and 10 items evaluating protective factors. The scores obtainable from the form range from 0 to 27. An increase in the score indicates a higher level of knowledge.
Care Skills | baseline (first assessment)
  The Sudden Infant Death Syndrome Care Skills Form was developed by the researchers based on the relevant literature to assess mothers' caregiving skills related to Sudden Infant Death Syndrome (SIDS). The form consists of 28 items and is designed as a 5-point Likert scale (Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree). The form consists of 28 items measuring the frequency of performing care skills. Participants rate each item on a scale from 'Always' (5 points) to 'Never' (1 point). Total scores range from 28 to 140. An increase in the score indicates that the individual performs care skills more frequently and regularly. Items with negative wording are reverse-scored.
Care Skills | 2 weeks after from baseline
  The Sudden Infant Death Syndrome Care Skills Form was developed by the researchers based on the relevant literature to assess mothers' caregiving skills related to Sudden Infant Death Syndrome (SIDS). The form consists of 28 items and is designed as a 5-point Likert scale (Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree). The form consists of 28 items measuring the frequency of performing care skills. Participants rate each item on a scale from 'Always' (5 points) to 'Never' (1 point). Total scores range from 28 to 140. An increase in the score indicates that the individual performs care skills more frequently and regularly. Items with negative wording are reverse-scored.
Care Skills | at the end of the invervention program (4 weeks after from baseline)
  The Sudden Infant Death Syndrome Care Skills Form was developed by the researchers based on the relevant literature to assess mothers' caregiving skills related to Sudden Infant Death Syndrome (SIDS). The form consists of 28 items and is designed as a 5-point Likert scale (Strongly Disagree, Disagree, Neutral, Agree, Strongly Agree). The form consists of 28 items measuring the frequency of performing care skills. Participants rate each item on a scale from 'Always' (5 points) to 'Never' (1 point). Total scores range from 28 to 140. An increase in the score indicates that the individual performs care skills more frequently and regularly. Items with negative wording are reverse-scored.
Self-Efficacy | baseline (first assessment)
  The General Self-Efficacy Scale is a five-point Likert-type scale. For each item, participants respond to the question "How well does this describe you?" using five options ranging from "Not at all" to "Very well." Each item is scored between 1 and 5. The scale consists of 17 items and demonstrates a three-factor structure: Initiation (9 items: 2, 4, 5, 6, 7, 10, 11, 12, 17), Perseverance (5 items: 3, 13, 14, 15, 16), and Sustained Effort (3 items: 1, 8, 9). The total score ranges from 17 to 85, with higher scores indicating greater self-efficacy.
Self-Efficacy | 2 weeks after from baseline
  The General Self-Efficacy Scale is a five-point Likert-type scale. For each item, participants respond to the question "How well does this describe you?" using five options ranging from "Not at all" to "Very well." Each item is scored between 1 and 5. The scale consists of 17 items and demonstrates a three-factor structure: Initiation (9 items: 2, 4, 5, 6, 7, 10, 11, 12, 17), Perseverance (5 items: 3, 13, 14, 15, 16), and Sustained Effort (3 items: 1, 8, 9). The total score ranges from 17 to 85, with higher scores indicating greater self-efficacy.
Self-Efficacy | at the end of the invervention program (4 weeks after from baseline)
  The General Self-Efficacy Scale is a five-point Likert-type scale. For each item, participants respond to the question "How well does this describe you?" using five options ranging from "Not at all" to "Very well." Each item is scored between 1 and 5. The scale consists of 17 items and demonstrates a three-factor structure: Initiation (9 items: 2, 4, 5, 6, 7, 10, 11, 12, 17), Perseverance (5 items: 3, 13, 14, 15, 16), and Sustained Effort (3 items: 1, 8, 9). The total score ranges from 17 to 85, with higher scores indicating greater self-efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared on request